CLINICAL TRIAL: NCT07014280
Title: Efficacy of Intralesional Bevacizumab Versus Intralesional Triamcinolone Acetonide Injection in the Treatment of Keloids.
Brief Title: Bevacizumab Versus Triamcinolone Acetonide for the Treatment of Keloids.
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Rana F Hilal, MD, Assistant professor, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BevaVSsteroid:keloids
Record Dates: First submitted 2025-05-16; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Keloids
MeSH Terms: conditions — Keloid | interventions — Bevacizumab; Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intralesional bevacizumab injection (Active Comparator): Intralesional bevacizumab injection for the treatment of keloid
  Interventions: Drug: Bevacizumab
- Intralesional corticosteroid injection (Active Comparator): Intralesional triamcinolone acetonide injection for the treatment of keloids
  Interventions: Drug: Triamcinolone Acetonide

INTERVENTIONS:
Drug: Bevacizumab — anti-VEGF
  Arms: Intralesional bevacizumab injection
Drug: Triamcinolone Acetonide — corticosteroid
  Arms: Intralesional corticosteroid injection

SUMMARY:
The study compares the efficacy and safety of intralesional bevacizumab versus corticosteroids for the treatment of keloids. Assessment will be done clinically by the use of Modified Vancouver Scar Scale. Erythema index will be measured by spectrophotometry. The levels of Vascular Endothelial Growth Factor, collagen type 1 and collagen type 3 in the lesions before and after each treatment modality.

ELIGIBILITY:
Inclusion Criteria:

* Patients with keloids (post-traumatic, any site, any duration)
* Age >18 years
* Patients who didn't receive any treatment for the lesions in the past 6 weeks

Exclusion Criteria:

* Patients who are pregnant, willing to get pregnant or lactating
* History of any liver or renal disease
* History of any cardiovascular disease
* History of hypertension
* History of thrombo-embolic events
* Known cases of bleeding disorders
* History of peptic ulcer
* Patients who underwent any surgeries in the last month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Modified Vancouver scar scale (mVSS) | 6 months
  Six characteristics of the scar were assessed. These are: vascularity, height, pliability, and pigmentation, pain and pruritis. Each characteristic is given a score, which are added together to give an overall score between 0 and 18. Higher scores mean a worse outcome.
Erythema Index | 6 months
  Evaluation of skin erythema index was done using a spectrophotometry device
Vascular Endothelial growth factor (VEGF) | 6 months
  Tissue levels of VEGF, collagen type 1 and 3 measured by Enzyme linked immunosorbent assay
Collagen type 1 and 3 | 6 months
  Tissue levels of collagen type 1 and 3 measured by Enzyme linked immunosorbent assay
Histopathological examination | 6 months
  Two mm punch biopsies were obtained per area at baseline and one month after the last treatment session. The post-treatment biopsy 3as taken from the vicinity of the baseline biopsy. Tissues are fixed in 10% buffered formalin, embedded in paraffin and sectioned into 5 μm-thick sections. Specimens were stained with hematoxylin and eosin (H&E) and orcein (or demonstration of elastic fibers). Histological examination was carried out under a light microscopy. Assessment was done as follows:
  1. Assessment of the collagen fibers will be done by examining H & E slides, putting grading from 1 to 4 according to the thickness and orientation of the collagen fibers and the spaces in between the fibers.
  2. Assessment of the elastic fibers will be done through examining orcein stained specimens and grading the elastic fibers in the scars from 1 to 4 based on presence or absence of the elastic fiber and degree of degradation and fragmentation.

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr El Ainy University Hospital, faculty of medicine, Cairo university, Cairo, El Manial, Egypt

IPD SHARING:
Plan to Share IPD: No